CLINICAL TRIAL: NCT05002218
Title: The Neural Effects of Balance Versus Aerobic Training in Individuals With Degenerative Cerebellar Diseases
Brief Title: Training in Ataxia - Individuals With Degenerative Cerebellar Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Scott Barbuto, Assistant Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAT8388; 1K23NS121518-01A1 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Cerebellar Ataxia
Keywords: ataxia; cerebellar ataxia; exercise; training; rehabilitation
MeSH Terms: conditions — Cerebellar Ataxia; Ataxia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single-blinded randomized control trial.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers and outcome assessor will not know which group individuals are assigned. In addition, the primary outcome will be video-recorded and the videos will be scrambled so that outcome assessor will not know if the test was done pre- or post-training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Training (Experimental): Participants will be given a stationary exercise bike for home use. They will be instructed to use the exercise bike five times a week for thirty-minute sessions. The exercise intensity prescription will be based on the subject's VO2max determined on pre-test day. The exercise program will start at 60% of intensity per session, and then will be increased by steps of 5% intensity every 2 sessions until participants reach 30 minutes of training at 80% intensity. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be instructed to log each training session. Subjects will record duration of exercise, perceived exertion, average heart rate, maximum heart rate, and distance.
  Interventions: Behavioral: Aerobic Training
- Balance Training (Active Comparator): A physical therapist will tailor a home balance training program for each participant based on pre- training capabilities. Subjects will be asked to perform exercises five times a week for thirty-minute sessions. Both dynamic and static exercises will be performed in sitting and standing positions. Exercises will start with stabilizing in a challenging static position and progress to dynamic arm and leg movements in the same or modified position. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be required to log their exercise effort in terms of frequency and level of balance challenge.
  Interventions: Behavioral: Balance Training

INTERVENTIONS:
Behavioral: Aerobic Training — Aerobic training on stationary bike 5x a week for 30 minutes a day.
  Arms: Aerobic Training
Behavioral: Balance Training — Balance training 5x a week for 30 minutes as instructed by a therapist. Standard of care.
  Arms: Balance Training

SUMMARY:
Balance and aerobic training show promise as treatments for degenerative cerebellar diseases, but the neural effects of both training methods are unknown. The goal of this project is to evaluate how each training method impacts the brain, and particularly, the degenerating cerebellum. Various neuroimaging techniques will be used to accomplish this goal and test the hypothesis that balance training impacts brain structures outside the cerebellum whereas aerobic training causes more neuroplastic changes within the cerebellum.

DETAILED DESCRIPTION:
Degenerative cerebellar diseases are a group of disorders that cause severe disability and can be fatal. There are currently no known disease-modifying treatments available for use, and there is a critical need to find treatments that slow disease progression and allow affected individuals to live more functional lives. Balance and aerobic training show promise as treatments for degenerative cerebellar diseases, but the neural effects of both training methods have not been thoroughly investigated. It is crucial to understand how the training impacts the brain, and particularly the cerebellum, in order to determine if one training method is better at slowing disease progression than the other. The goal of this proposal is to compare the neural effects of balance versus aerobic training in individuals with degenerative cerebellar diseases. The investigator hypothesizes that aerobic training causes neuroplastic changes within the cerebellum whereas balance training causes improvements for people with cerebellar degeneration by impacting brain structures outside the cerebellum. If this hypothesis is true, aerobic training may have more influence on disease progression than balance training as it directly impacts the cerebellum.

To investigate the hypothesis, various neuroimaging techniques will be used. In AIM 1, the investigator will compare cerebellar volume before and after the participants perform either 6-months of balance or aerobic training. In AIM 2, the investigator will investigate whether neural changes have clinical significance by correlating cerebellar volume changes with clinical measures of ataxia. Finally, for AIM 3, the investigator will use diffusion tensor imaging and resting state fMRI scans to examine how both training methods impact cerebellar microstructure and functional cerebellar connections. The investigator hopes that a detailed understanding of how each training method impacts the cerebellum will lead to more targeted training regimens with the goal of slowing disease progression of these devastating diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spinocerebellar ataxia
* Cerebellar atrophy on MRI
* Prevalence of ataxia on clinical exam
* Ability to safely ride a stationary exercise bike

Exclusion Criteria:

* Other neurologic conditions
* Heart disease
* Cognitive impairment
* Medical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Barbuto, MD, Principal Investigator — Assistant Professor of Rehabilitation and Regenerative Medicine
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barbuto S, Lee S, Stein J, Kuo SH, Quinn L, Spinner M, Stern Y. Home Training for Cerebellar Ataxias: A Randomized Clinical Trial. JAMA Neurol. 2025 Nov 1;82(11):1162-1170. doi: 10.1001/jamaneurol.2025.3421. PMID 40946705

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 64 participants were enrolled. Of those, 2 participants withdrew from the study prior to randomization.
Period: Overall Study
Arm/Group | Aerobic Training | Balance Training
Started | 31 | 31
Completed | 26 | 25
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Training | Balance Training | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (12.5) | 53.8 (13.5) | 54.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 15 | 18 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 31 | 62
Disease duration [Mean (Standard Deviation); unit: years] | 8.2 (7.0) | 6.8 (6.8) | 7.6 (6.9)
Disease type [Count of Participants; unit: Participants]
  Spinocerebellar ataxia type 1 (SCA1) | 2 | 5 | 7
  SCA2 | 5 | 4 | 9
  SCA3 | 4 | 2 | 6
  SCA4 | 1 | 1 | 2
  SCA6 | 5 | 3 | 8
  SCA7 | 0 | 1 | 1
  SCA8 | 2 | 4 | 6
  SCA14 | 1 | 0 | 1
  SCA15 | 1 | 0 | 1
  SCA19 | 0 | 1 | 1
  SCA27 | 0 | 1 | 1
  Idiopathic | 8 | 9 | 17
  multiple system atrophy-cerebellar type | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Assessment and Rating of Ataxia (SARA) Score
Description: This is to measure ataxia severity. The Scale for the Assessment and Rating of Ataxia (SARA) will be administered before and after training. SARA is an 8-item performance based scale, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia) - with higher scores indicating more severe ataxia. The scores are based on patient performance of gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movements and heel-shin slide. The change in score from baseline to 6 months, 9 months, and 12 months will be reported.
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: Some participants were lost to follow up at 6 months, 9 months, and 12 months, so data could not be collected from those participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline to 6 months: number analyzed (Participants) | 29 | 27
  Baseline to 6 months | -2.4 [-3.1 to -1.8] | -0.9 [-1.5 to -0.2]
  Baseline to 9 months: number analyzed (Participants) | 27 | 25
  Baseline to 9 months | -1.5 [-2.2 to -0.8] | -0.2 [-0.84 to 0.5]
  Baseline to 12 months: number analyzed (Participants) | 26 | 25
  Baseline to 12 months | -1.4 [-2.1 to -0.7] | 0 [-0.66 to 0.70]

2. Secondary Outcome: Average Gait Speed
Description: This is to measure average time to complete 8-meter walk test. Participants will walk 8 meters as fast as possible three different times. Gait will be reported as meters per second (m/s).
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
m/s
  Baseline | 0.90 (0.28) | 0.95 (0.32)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 0.80 (0.26) | 0.89 (0.30)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 0.80 (0.26) | 0.80 (0.26)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 0.80 (0.26) | 0.79 (0.26)

3. Secondary Outcome: Dynamic Gait Index Score
Description: The dynamic gait index (DGI) will be performed to assess balance. Patients will be asked to walk 20 feet and conditions such as speed and head position will be varied as previously described. The examiner will then grade the subject's movement on a four-point ordinal scale, ranging from 0 (lowest level of function) to 3 (highest level of function). The total score range is 0 to 24, with higher scores indicating better dynamic balance and functional mobility.
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline | 11.8 (2.0) | 11.7 (2.0)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 12.8 (2.0) | 13.2 (2.0)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 13.0 (2.0) | 13.2 (2.0)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 13.3 (2.0) | 12.8 (2.0)

4. Secondary Outcome: Timed Up and Go (TUG)
Description: The Timed Up and Go will be performed to assess balance. Once the tester says "Go", participants will stand from seated and walk around a cone that is 3 meters away, then walk back to the chair and sit back down. Participants will be timed from the moment the tester says "Go" until seated again.
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
seconds
  Baseline | 17.0 (3.1) | 16.6 (3.1)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 15.5 (3.1) | 15.7 (3.1)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 15.5 (3.1) | 15.7 (3.1)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 16.8 (3.1) | 16.7 (3.1)

5. Secondary Outcome: Fatigue Severity Scale (FSS) Score
Description: The FSS is a nine-item questionnaire that measures the severity of fatigue. Each item is rated on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree). Scores for all nine items are summed to calculate the total score, which ranges from 9 to 63. Higher scores indicate greater fatigue severity.
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline | 41.2 (5.1) | 33.5 (5.2)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 33.3 (5.2) | 35.0 (5.1)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 35.6 (5.2) | 34.8 (5.2)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 35.3 (5.2) | 36.2 (5.2)

6. Secondary Outcome: Quality of Life (QOL) - Physical Health
Description: The WHOQOL-BREF measures self-perceived quality of life across four domains: Physical Health, Psychological, Social Relationships, and Environment. Scores are derived from a 5-point Likert scale, with higher scores indicating better quality of life in that specific area. To calculate the domain scores, the mean score for items within each domain is multiplied by 4, and these scores are transformed to a 0 - 100 scale for interpretation.
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline | 55.8 (7.0) | 59.1 (7.1)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 54.3 (7.1) | 60.1 (7.1)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 57.1 (7.1) | 59.8 (7.2)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 57.1 (7.1) | 60.7 (7.2)

7. Secondary Outcome: Quality of Life (QOL) - Psychological
Description: as for outcome 6
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline | 65.6 (7.1) | 68.1 (7.2)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 63.1 (7.2) | 67.6 (7.2)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 68.8 (7.2) | 67.0 (7.2)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 66.2 (7.2) | 66.2 (7.2)

8. Secondary Outcome: Quality of Life (QOL) - Social Relationships
Description: as for outcome 6
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline | 60.1 (8.4) | 64.8 (8.5)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 65.5 (8.4) | 53.0 (8.4)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 64.2 (8.5) | 60.1 (8.5)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 65.4 (8.6) | 65.7 (8.5)

9. Secondary Outcome: Quality of Life (QOL) - Environment
Description: as for outcome 6
Time Frame: Baseline, 6 months, 9 months, 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aerobic Training | Balance Training
Number analyzed (Participants) | 31 | 31
score on a scale
  Baseline | 65.5 (5.7) | 68.3 (5.7)
  6 months: number analyzed (Participants) | 29 | 27
  6 months | 70.5 (5.7) | 66.1 (5.7)
  9 months: number analyzed (Participants) | 27 | 25
  9 months | 69.5 (5.7) | 69.6 (5.7)
  12 months: number analyzed (Participants) | 26 | 25
  12 months | 68.9 (5.7) | 72.2 (5.7)

10. Secondary Outcome: Prevalence of Desired Changes in Diffuse Tensor Imaging
Description: Diffusion data will be preprocessed for motion and corrected for geometrical distortion using ExploreDTI. For each participant, the bmatrix will be reoriented to provide a more accurate estimate of diffusion tensor orientations. Diffusion tensor estimation will be performed using a non-linear least square fitting method. FA and Mean Diffusivity (MD) maps will be generated. Whole brain tractography will be performed using all brain voxels with FA ≤ 0.2 as seed region.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2026-10

11. Secondary Outcome: Prevalence of Cerebellar Volume
Description: To determine cerebellar volume, each T1 scan will be visually inspected to ensure inclusion of only minimal movement artifacts. All images will be processed in a blinded manner in order to maintain accuracy and consistency of volume calculation. Regional cerebellar volumes will be calculated using the SUIT toolbox of the SPM12 software.
Time Frame: Baseline, 6 months, 9 months, 12 months
Reporting Status: Not Posted, anticipated posting 2026-10

12. Secondary Outcome: Prevalence of Desired Changes in Resting State fMRI Scans
Description: This measure will be a primary outcome for Aim 3. The anatomical and functional data will be pre-processed and analyzed using Statistical Parametric Mapping (SPM12) and the CONN toolbox Version 14p.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2026-10

ADVERSE EVENTS:
Time Frame: AE data was collected during in-person assessments at baseline, 6 months, 9 months, and 12 months
Arm/Group | Aerobic Training | Balance Training
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/31 | 1/31
Other Adverse Events (participants affected / at risk) | 8/31 | 10/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Training (N=31) | Balance Training (N=31)
Infection, hospitalized (Infections and infestations) | 0 | 1
Car Accident, hospitalized (Social circumstances) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Training (N=31) | Balance Training (N=31)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Falls (General disorders) | 2 | 8
Fatigue (General disorders) | 2 | 1
Infection, not hospitalized (Infections and infestations) | 4 | 4

LIMITATIONS AND CAVEATS:
The study had a small sample size and was conducted during the COVID-19 pandemic, precluding cardiopulmonary exercise testing. Recruitment was largely limited to individuals with multiple system atrophy-cerebellar type and idiopathic cerebellar ataxia, as individuals with other types of ataxia were recruited for other competing trials. Training adherence relied on training logs with no objective measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05002218/Prot_SAP_000.pdf